CLINICAL TRIAL: NCT01661699
Title: Oxidative Stress in Obstructive Sleep Apnea: Correlation of Biomarkers and Nasal CPAP Compliance
Status: Completed | Type: Observational
Sponsor: Georgetown University (Other)
Responsible Party: Principal Investigator, Christina Reichner, M.D., M.D., Associate Professor Medicine, Georgetown University
Other Study IDs: 2011-416
Record Dates: First submitted 2012-08-03; First posted 2012-08-09 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleep apnea: Those suspected of sleep apnea and scheduled for polysomnography and treated with CPAP therapy.

SUMMARY:
The purpose of this study is to check blood and urine levels to further define markers/tests in the blood and urine that would be useful in following patients with obstructive sleep apnea and then to see if by wearing CPAP every night, these markers can be reduced. This research is being done because currently there are no effective blood or urine markers to determine how well CPAP is working.

DETAILED DESCRIPTION:
The goal of this study is to further define biomarkers that would be useful in following patients with obstructive sleep apnea and examining their response to compliance to therapy with CPAP. To date no correlation between biomarkers of oxidative stress and compliance to CPAP has been measured. CPAP is the most effective treatment for obstructive sleep apnea and has been show to reduce blood pressure and decrease oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women over 18 years suspected of having sleep apnea

Exclusion Criteria:

* Those under 18 years or not suspected of having sleep apnea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Those over 18 years suspected of having sleep apnea.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Determining biomarkers for polysomnography characteristics before and after CPAP treatment | 6 months
  The primary objective of this pilot study will determine the biomarkers for polysomnography characteristics with CPAP treatment from baseline to 6 months in patients with obstructive sleep apnea. The results will guide biomarker selection for full scale studies.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Reichner, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Hospital, Washington D.C., District of Columbia, United States